CLINICAL TRIAL: NCT00003264
Title: Phase II Evaluation of Weekly Cisplatin and Gemcitabine in the Treatment of Advanced (Recurrent or Metastatic) Carcinoma of the Head and Neck
Brief Title: Cisplatin Plus Gemcitabine in Treating Patients With Advanced Squamous Cell Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066159; P30CA006927 (NIH); FCCC-97021 (Other: Fox Chase Cancer Center); NCI-G98-1403 (Other: National Cancer Institute)
Record Dates: First submitted 1999-11-01; First posted 2004-03-01 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Head and Neck Cancer
Keywords: stage IV salivary gland cancer; recurrent salivary gland cancer; recurrent metastatic squamous neck cancer with occult primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma; salivary gland squamous cell carcinoma; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of cisplatin plus gemcitabine in treating patients with advanced squamous cell head and neck cancer that cannot be treated by surgery or radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the response rate and toxicity of weekly cisplatin and gemcitabine in patients with recurrent or metastatic squamous cell carcinoma of the head and neck who have received either no prior chemotherapy or no more than one prior chemotherapy regimen for advanced disease.

OUTLINE: Patients are stratified according to prior chemotherapy status: chemotherapy naive (no prior chemotherapy, or prior neoadjuvant or adjuvant chemotherapy at least 6 months prior to recurrence, or prior biologic agents only) vs chemotherapy exposed (one prior chemotherapy regimen directed at recurrent or newly diagnosed metastatic disease and/or prior neoadjuvant or adjuvant chemotherapy less than 6 months prior to recurrence). Patients receive gemcitabine as a 30 minute infusion weekly for 3 weeks followed by one week of rest. Cisplatin is administered as a 30-60 minute infusion immediately preceding gemcitabine. Treatment repeats every 28 days for 2-6 courses, depending on response. Patients with previously untreated metastatic disease may have treatment interrupted to receive radiation therapy to locoregional disease sites. Patients may continue treatment beyond 6 courses at the discretion of the physician. Patients are followed every 3 months.

PROJECTED ACCRUAL: This study will accrue approximately 36 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven squamous cell carcinoma of the head and neck considered incurable with surgery or radiation therapy Bidimensionally measurable disease or readily evaluable disease by either physical exam or radiography Biopsy proven recurrence following completion of radiotherapy required if only site of measurable disease is within a previous radiation port

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 2000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Neurologic: Peripheral sensory neuropathy no greater than grade 1 Other: No significant active infection (patients with WBC of 12,000/mm3 or greater, or fever of 100.6 degrees F or higher, must be evaluated to rule out occult infection) Not pregnant or nursing Effective contraception required of fertile patients No active second malignancy

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior biologic therapy (interleukin-2, interferon, monoclonal antibodies, and/or retinoids) permitted Recovered from prior biologic therapy Chemotherapy: No more than one prior chemotherapy regimen for advanced or relapsed disease No chemotherapy within 4 weeks prior to study Prior neoadjuvant or radiosensitizing chemotherapy allowed Endocrine therapy: Not specified Radiotherapy: Prior radiotherapy permitted Recovered from prior radiotherapy Surgery: Recovered from major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 1997-10; Primary Completion 2002-02 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey J. Langer, MD, Study Chair — Fox Chase Cancer Center
Locations (12):
- United States (12):
  - Hunterdon Regional Cancer Center, Flemington, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Riverview Medical Center - Booker Cancer Center, Red Bank, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - St. Luke's Network - Bethlehem, Bethlehem, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Harrisburg Polyclinic Medical Center, Harrisburg, Pennsylvania
  - Saint Mary Regional Center, Langhorne, Pennsylvania
  - North Penn Hospital, Lansdale, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania